CLINICAL TRIAL: NCT05908916
Title: A Single-arm Phase II Trial of Atezolizumab and Bevacizumab With Combined Radiotherapy in Advanced Hepatocellular Carcinoma With Portal Vein Invasion
Brief Title: Atezolizumab and Bevacizumab With Combined Radiotherapy for Advanced Hepatocellular Carcinoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4-2023-0384
Record Dates: First submitted 2023-06-09; First posted 2023-06-18 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Therapeutic arm (Experimental): AtezoBev with combined radiotherapy
  Interventions: Drug: AtezoBev with combined radiotherapy

INTERVENTIONS:
Drug: AtezoBev with combined radiotherapy — Atezolizumab (1200mg) and Bevacizumab (15mg/kg) are administered to patients once for each cycle with 3-week intervals, and additional radiotherapy (iGTV 50-60 Gy, CTV 40Gy, PTV 30Gy / 10Fx) for the mass or portal vein tumor thrombosis is performed before second cycle of AtezoBev.

SUMMARY:
Atezolizumab plus Bevacizumab combination therapy (AtezoBev) is well-known 1st-line therapy for advanced hepatocellular carcinoma (HCC). However, there are unmet needs for patients with advanced HCC who do not respond to AtezoBev. External beam radiotherapy (RT) is another well-known locoregional therapy for HCC that induces inflammatory cascade and abscopal effect as a systemic anticancer effect and enhances the effect of AtezoBev. Therefore, the investigators aim to verify the effect of AtezoBev plus RT for advanced HCC through this single-center, prospective phase II one-armed cohort study over three years. This study recruits 51 patients to verify the effect of the intervention. Atezolizumab (1200mg) and Bevacizumab (15mg/kg) are administered to patients once for each cycle at 3-week intervals, and additional radiotherapy for the mass or portal vein tumor thrombosis is performed before second cycle of AtezoBev. The primary endpoint is progression-free survival by using response evaluation with modified RECIST.

ELIGIBILITY:
Inclusion Criteria:

1. age ≥19;
2. clinically or histologically diagnosed HCC;
3. HCC with Vp2-Vp4 portal vein invasion;
4. intact liver function with Child-Pugh class A;
5. adequate size of RT field;
6. intact performance with ECOG below 2;
7. non-pregnant with acceptable contraception in premenopausal women);
8. without other life-threatening diseases;
9. ability to provide written informed consent and to comply with all study conditions.

Exclusion Criteria:

1. Active uncontrolled infection;
2. Current or history (< or = 5 years) of advanced malignancies in the other organs;
3. History of liver transplantation;
4. miliary HCC which incompatible external beam RT

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Estimated)
Dates: Start 2023-07 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 2 years (per 9 weeks)
  Duration between AtezoBev initiation and tumor progression by mRECIST or patient's death

CONTACTS AND LOCATIONS:
Overall Officials: Do Young Kim, Principal Investigator — Severance Hospital
Locations (1):
- Severance hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No